CLINICAL TRIAL: NCT04593511
Title: An Open-Label Study in Healthy Volunteers to Evaluate the Safety, Tolerability and Pharmacokinetics of Four Formulations of LY03009 After a Single Intramuscular Injection
Brief Title: to Evaluate the Safety, Tolerability and Pharmacokinetics of Four Formulations of LY03009 in Healthy Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Luye Pharma Group Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LY03009/CT-AUS-101
Record Dates: First submitted 2020-09-21; First posted 2020-10-20 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Formulation 1 (Experimental): a single dose of LY03009 F1
  Interventions: Drug: LY03009 F1
- Formulation 2 (Experimental): a single dose of LY03009 F2
  Interventions: Drug: LY03009 F2
- Formulation 3 (Experimental): a single dose of LY03009 F3
  Interventions: Drug: LY03009 F3
- Formulation 4 (Experimental): a single dose of LY03009 F4
  Interventions: Drug: LY03009 F4

INTERVENTIONS:
Drug: LY03009 F1 — a single dose of LY03009 F1
  Arms: Formulation 1
Drug: LY03009 F2 — a single dose of LY03009 F2
  Arms: Formulation 2
Drug: LY03009 F3 — a single dose of LY03009 F3
  Arms: Formulation 3
Drug: LY03009 F4 — a single dose of LY03009 F4
  Arms: Formulation 4

SUMMARY:
The purpose of this study is to Evaluate the Safety, Tolerability and Pharmacokinetics of Four Formulations of LY03009 in Healthy Volunteers.

DETAILED DESCRIPTION:
This is an open-label study in healthy volunteers to evaluate the safety, tolerability and pharmacokinetics of four formulations of LY03009 (F1, F2, F3, F4) after a single intramuscular injection.

Approximately 40 healthy subjects are planned to be enrolled in this study and assigned to four cohorts (F1, F2, F3, F4) sequentially, 10 subjects per group at a fixed dose of 112 mg for F1~F3 and 224 mg for F4. Each subject will receive only one dose in this study.

ELIGIBILITY:
Inclusion Criteria：

To participate in the study, subjects must meet all of the following inclusion criteria:

1. Willing and capable of giving signed written informed consent;
2. Male or female, 18-65 years of age (inclusive) at screening;
3. Body mass index (BMI, weight [kg]/height [m]2) between 18.0 and 30.0 kg/m2, inclusive;
4. The screening results within the normal range or outside the normal range but assessed as clinically non-significant by the Investigator based on detailed medical history, clinical laboratory tests, vital signs, physical examination, and 12-lead ECG; QTcF ≤450 msec for male subjects, and QTcF ≤470 msec for female subjects.
5. Males who are willing to remain abstinent; or if engaging in sexual intercourse with a female partner of childbearing potential, willing to use a condom in addition to having the female partner use a highly effective method of contraception throughout the study and until at least 3 months after the end of the study. This requirement does not apply to subjects in a same sex relationship or subjects with female partners of non-childbearing potential. Male subjects must also be willing to not donate sperm throughout the study and until at least 3 months after the end of the study.

Exclusion Criteria：

Subjects meeting any of the following criteria will be excluded from the study:

1. With history of history of gastrointestinal, cardiovascular, musculoskeletal, endocrine, hematologic, psychiatric, renal, hepatic, neurologic, bronchopulmonary, immunologic, and/or lipid metabolism disorders, and/or drug hypersensitivity, or any other condition that, in the opinion of the PI, would jeopardize the safety of the subject, affect the validity of the study results, or impair the ability to provide informed consent;
2. Hospital admission or major surgery within 3 months prior to screening, or plan to have surgery before the completion of study;
3. Receipt of another investigational product within 1 month or 5 half-lives of the other investigational product, whichever is longer, before study drug administration in this study;
4. Unwillingness or inability to comply with food and beverage restrictions during study participation;
5. Have a history of significant drug sensitivity or drug allergy, or known hypersensitivity to the study drugs, the metabolite or formulation excipients;
6. Malignancy within 5 years of screening visit (excluding non-melanoma skin cancer and cervical carcinoma in situ that has been completely resected);
7. Subject who is considered unsuitable for participating in the study in the opinion of investigator.
8. Recent administration of live vaccine within 3 months prior to dosing and until at least 30 days after the completion of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-02-02 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Frequency of adverse events | From screening up to day 98
  Frequency of adverse events. Apply to cohort F1, cohort F2 and cohort F3.
Frequency of adverse events | From screening up to day 161
  Frequency of adverse events. Apply to cohort F4.

SECONDARY OUTCOMES:
Maximum (peak) plasma concentration (Cmax) of LY03009 | From screening up to day 98
  Maximum (peak) plasma concentration (Cmax) of LY03009. Apply to cohort F1, cohort F2 and cohort F3.
Maximum (peak) plasma concentration (Cmax) of LY03009 | From screening up to day 161
  Maximum (peak) plasma concentration (Cmax) of LY03009. Apply to cohort F4
Area under the plasma concentration-time curve from time zero to the last measurable concentration (AUC0-t) of LY03009 | From screening up to day 98
  Area under the plasma concentration-time curve from time zero to the last measurable concentration (AUC0-t) of LY03009.Apply to cohort F1, cohort F2 and cohort F3.
Area under the plasma concentration-time curve from time zero to the last measurable concentration (AUC0-t) of LY03009 | From screening up to day 161
  Area under the plasma concentration-time curve from time zero to the last measurable concentration (AUC0-t) of LY03009.Apply to cohort F4
Area under the plasma concentration-time curve from time zero to infinity (AUC0-∞) of LY03009 | From screening up to day 98
  Area under the plasma concentration-time curve from time zero to infinity (AUC0-∞) of LY03009.Apply to cohort F1, cohort F2 and cohort F3.
Area under the plasma concentration-time curve from time zero to infinity (AUC0-∞) of LY03009 | From screening up to day 161
  Area under the plasma concentration-time curve from time zero to infinity (AUC0-∞) of LY03009. Apply to cohort F4
Time to maximum plasma concentration (Tmax) of LY03009 | From screening up to day 98
  Time to maximum plasma concentration (Tmax) of LY03009. Apply to cohort F1, cohort F2 and cohort F3.
Time to maximum plasma concentration (Tmax) of LY03009 | From screening up to day 161
  Time to maximum plasma concentration (Tmax) of LY03009. Apply to cohort F4
Terminal elimination half-life (t1/2) of LY03009 | From screening up to day 98
  Terminal elimination half-life (t1/2) of LY03009. Apply to cohort F1, cohort F2 and cohort F3.
Terminal elimination half-life (t1/2) of LY03009 | From screening up to day 161
  Terminal elimination half-life (t1/2) of LY03009.Apply to cohort F4
Apparent clearance (CL/F) of LY03009 | From screening up to day 98
  Apparent clearance (CL/F) of LY03009. Apply to cohort F1, cohort F2 and cohort F3.
Apparent clearance (CL/F) of LY03009 | From screening up to day 161
  Apparent clearance (CL/F) of LY03009. Apply to cohort F4
Apparent volume of distribution (Vz/F) of LY03009 | From screening up to day 98
  Apparent volume of distribution (Vz/F) of LY03009. Apply to cohort F1, cohort F2 and cohort F3.
Apparent volume of distribution (Vz/F) of LY03009 | From screening up to day 161
  Apparent volume of distribution (Vz/F) of LY03009. Apply to cohort F4
Terminal elimination rate constant (λz) of LY03009 | From screening up to day 98
  Terminal elimination rate constant (λz) of LY03009. Apply to cohort F1, cohort F2 and cohort F3.
Terminal elimination rate constant (λz) of LY03009 | From screening up to day 161
  Terminal elimination rate constant (λz) of LY03009. Apply to cohort F4
Mean residence time (MRT) of LY03009 | From screening up to day 98
  Mean residence time (MRT) of LY03009. Apply to cohort F1, cohort F2 and cohort F3.
Mean residence time (MRT) of LY03009 | From screening up to day 161
  Mean residence time (MRT) of LY03009. Apply to cohort F4
Area under the plasma concentration-time curve extrapolated from time t to infinity as a percentage of total AUC (%AUCex) of LY03009 | From screening up to day 98
  Area under the plasma concentration-time curve extrapolated from time t to infinity as a percentage of total AUC (%AUCex) of LY03009. Apply to cohort F1, cohort F2 and cohort F3.
Area under the plasma concentration-time curve extrapolated from time t to infinity as a percentage of total AUC (%AUCex) of LY03009 | From screening up to day 161
  Area under the plasma concentration-time curve extrapolated from time t to infinity as a percentage of total AUC (%AUCex) of LY03009. Apply to cohort F4

CONTACTS AND LOCATIONS:
Overall Officials: Angela Molga, Principal Investigator — CMAX Clinical Research Pty Ltd
Locations (1):
- CMAX clinical Research Pty Ltd, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No